CLINICAL TRIAL: NCT02588417
Title: Intrathecal Levobupivacaine Versus A Combination of Levobupivacaine and Dexamethasone in Parturients Receiving Combined Spinal Epidural for Vaginal Delivery Analgesia: A Comparative Study.
Brief Title: Intrathecal Dexamethasone and Labor Analgesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ahmed elsakka (Other)
Responsible Party: Sponsor-Investigator, ahmed elsakka, dr, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: no id
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Effects of; Anesthesia, in Labor and Delivery
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone (Active Comparator): dexamethasone 4 mg administered intrathecally during active stage of labor once only in combination with levobupivacaine
  Interventions: Drug: Dexamethasone; Drug: Levobupivacaine
- levobupivacaine (Active Comparator): levobupivacaine 2.5 mg in 2 ml administered intrathecally during active stage of labor once and alone and then epidural levobupivacaine 7ml of 2.5 mg concentrationis administered till the end of labor
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Dexamethasone — 4mg dexamethasone intrathecally plus levobupivacaine 2.5 mg
  Other Names: decadron
  Arms: dexamethasone
Drug: Levobupivacaine — levobupivacaine 2.5 mg
  Other Names: chirocaine

SUMMARY:
To evaluate the effectiveness of adding dexamethasone to intrathecal levobupivacaine in combined spinal epidural (CSE) analgesia during vaginal delivery.

DETAILED DESCRIPTION:
This prospective double-blind trial included 80 primigravidas during vaginal delivery with a cervical dilatation ≥ 4 cm and 50% effacement randomly assigned to one of two equal groups; Group L received intrathecal levobupivacaine 0.25% in 2 mL and Group LD received intrathecal levobupivacaine 0.25% combined with dexamethasone 4 mg in 2 mL. At first request of analgesia, a combination of 0.25% levobupivacaine with 100 μg fentanyl in 10 ml via the epidural catheter. Further analgesia was provided with 7 ml 0.25% levobupivacaine hourly. The primary outcome measure was the duration of spinal analgesia. Secondary outcome measures include time from spinal analgesia to delivery, total amount of epidurally administered levobupivicaine, adverse effects of neuraxial block and neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I,II patients schedueled for normal vaginal deliveries
* age between 18-35 years old

Exclusion Criteria:

* Patients who refused to participate
* complicated pregnancies

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
duration of spinal analgesia | 1 day

SECONDARY OUTCOMES:
time from spinal analgesia to delivery | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: nadia yo helmy, md, Principal Investigator — professor of anaesthesia cairo university